CLINICAL TRIAL: NCT00452569
Title: Randomised, Controlled, Open-labelled, Multi-centre Comparison of Thalidomide Versus High-dose Dexamethasone for the Treatment of Relapsed Refractory Multiple Myeloma
Brief Title: Efficacy and Safety Study of 3 Thalidomide Doses for the Treatment of Relapsed Refractory Multiple Myeloma
Acronym: OPTIMUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THA PH INT 2005 CL001
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): Oral thalidomide (100mg/day) administered to the patient once daily until progression of the disease and for a maximum of 336 +/- 36 days (12 cycles of 28 +/- 3 days).
  Interventions: Drug: Thalidomide
- B (Experimental): Oral thalidomide (200mg/day) administered to the patient once daily until progression of the disease and for a maximum of 336 +/- 36 days (12 cycles of 28 +/- 3 days).
  Interventions: Drug: Thalidomide
- C (Experimental): Oral thalidomide (400mg/day) administered to the patient once daily until progression of the disease and for a maximum of 336 +/- 36 days (12 cycles of 28 +/- 3 days).
  Interventions: Drug: Thalidomide
- D (Active Comparator): High dose oral dexamethasone will be administered at a dose of 40mg/day on days 1-4, 9-12 and 17-20 of each 28-day cycle for cycles 1-4. Beginning with cycle 5, the oral dexamethasone dosing schedule will be reduced to 40mg/day on days 1-4 of each 28-day cycle. Dexamethasone will be administered until progression of the disease and for a maximum of 336 +/- 36 days (12 cycles of 28 +/- 3 days).
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Thalidomide — Oral thalidomide (100mg or 200mg or 400 mg/day) administered to the patient once daily until progression of the disease and for a maximum of 336 + 36 days (12 cycles of 28 +/- 3 days).
  Arms: A; B; C
Drug: Dexamethasone — High dose oral dexamethasone will be administered at a dose of 40mg/day on days 1-4, 9-12 and 17-20 of each 28-day cycle for cycles 1-4. Beginning with cycle 5, the oral dexamethasone dosing schedule will be reduced to 40mg/day on days 1-4 of each 28-day cycle. Dexamethasone will be administered until progression of the disease and for a maximum of 336 +/- 36 days (12 cycles of 28 +/- 3 days).
  Arms: D

SUMMARY:
The primary objective is to compare the time to progression (TTP) of three daily doses of thalidomide (100, 200 and 400 mg) with high-dose dexamethasone in relapsed refractory multiple myeloma (MM) patients and to subsequently select the optimum thalidomide dose in terms of median TPP and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged ≥ 18 years at the time of signing the informed consent form
* Patients who have been previously diagnosed with MM who have received between 1 & 3 prior lines of treatment for their disease, and who require therapy because of disease progression
* Secretory MM with measurable levels of monoclonal protein in serum (> 10 g/L of IgG M-protein or > 5 g/L of IgA M-protein) or urine (≥ 200 mg/ 24hours); Patient with the following rare subclasses of the immunoglobulin: IgD, IgE, IgM can be included in the study if the level of monoclonal protein in serum is > 5g/L or ≥ 200 mg/24hours in urine. As IgM immunoglobulin isotype can be related to Waldenstrom's macroglobulinemia, it is important to distinguish and not include in the study patients with Waldenstrom's macroglobulinemia.
* ECOG performance status of 0, 1, or 2
* Life expectancy >3months
* Able to adhere to the study visit schedule & other protocol requirements
* Women of child-bearing potential must agree to use 2 methods of contraception for at least 4weeks before starting the therapy, during the Treatment Period, & for 4 weeks after the last dose
* Males must agree to use barrier contraception (latex condoms) when engaging in reproductive activity during the Treatment Period & for 4 weeks after the last dose
* Written, informed consent

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the Informed Consent Form
* Pregnant or lactating women. A serum β-hCG pregnancy test must be performed at the Screening visit for female patients of child-bearing potential. If the test is positive, the patient must be excluded from the study. Confirmation that the patient is not pregnant must be established by a negative serum or urinary pregnancy test with the result obtained 1day prior to the Baseline visit (or the day of the visit if results are available before drug delivery). A pregnancy test is not required for naturally post-menopausal women (who have not had menses at any time in the preceding 24 consecutive months) or surgically sterilized women (hysterectomy, bilateral ovariectomy, bilateral salpingectomy)
* Non-secretory MM
* Any of the following laboratory abnormalities: Absolute neutrophil count (ANC) <500 cells/mm3 (0.5 x 109/L); Platelet count <30,000/mm3 (30.0 x 109L) without transfusion support within 7 days before the test; Serum creatinine >3.0mg/dL (265μmol/L); Serum aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) >3.0 x upper limit of normal (ULN); Serum total bilirubin >2.0mg/dL (34μmol/L)
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if s/he were to participate in the study, or which confounds the ability to interpret data from the study
* Severe cardiac dysfunction (according to the New York Heart Association [NYHA] classification III-IV)
* Severe bradycardia (<50bpm)
* Peripheral neuropathy ≥Grade 2 in severity (according to the NCI CTC Version 3.0)
* Prior history of malignancy (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the patient has been free of disease for ≥5years
* Patient received any chemotherapy, corticosteroids (> 10 mg/day prednisone or equivalent as a continuous dose) within 4 weeks before randomization
* Previously treated with thalidomide or thalidomide derivatives
* Patients refractory to high-dose dexamethasone (defined as experiencing less than a PR to dexamethasone, or PD within 6months after discontinuing dexamethasone, or discontinued dexamethasone because of ≥Grade 3 dexamethasone-related toxicity. Previous high-dose dexamethasone therapy is defined as >500mg dexamethasone or equivalent over a 10week period, whether administered alone or as part of the VAD regimen)
* Contraindications for high-dose dexamethasone
* Active or chronic gastrointestinal ulcers, active viral infections (herpes, varicella, HIV, hepatitis B, hepatitis C), glaucoma, uncontrolled hypertension, or diabetes mellitus, unless well controlled & under strict supervision during dexamethasone treatment
* Patient enrolled in another clinical trial or who have participated in another trial with the last 4weeks before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2006-02-01 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2009-01-01 (Actual)

PRIMARY OUTCOMES:
The evaluation of Independent Review Committee-documented time to progression (TTP). | >160 "IRC confirmed" disease progression in the Dexamethasone or Thalidomide 400 mg/day arms

SECONDARY OUTCOMES:
Response rate (CR + PR), according to the EBMT criteria | Every 4 weeks
Response duration | Every 4 weeks
Clinical benefit as measured by ECOG performance status, transfusion requirement and Grade ≥3 infections (assessed by the National Cancer Institute Common Toxicity Criteria) | Every 4 weeks
Progression-free survival (PFS) | Disease progression evaluated every 4 weeks
Overall survival (OS) | Evaluated after 150 deaths occurring in Dexamethasone and Thalidomide 400 mg arms
Composite of disease progression and death (recurrent time(s) from randomisation to disease progression and/or death) | Evaluated after 160 "IRC confirmed" disease progression in the Dexamethasone or Thalidomide 400 mg/day arms
Quality of life as determined by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) | Baseline/Week 8/ Week 16/Week 24/Week 32/Week 40/Week 48
Adverse events (AEs) | Every 4 weeks
Assessment of peripheral neuropathy | Screening, Week 24, Week 48
Vital signs and physical examination | Every 4 weeks
Clinical laboratory tests | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kropff, MD, Principal Investigator — Universitatsklinikum Munster
Locations (86):
- Bulgaria (6):
  - Clinic of Haematology, University Multiprofiled Hospital for Active Treatment "G. Stranski", Pleven
  - Clinic of Haematology, University Multiprofiled Hospital for Active Treatment, Plovdiv
  - University of Multiprofiled Hospital for Active Treatment "Alexandrovska" - Sofia, Sofia
  - Military Medical Academy/Dept Haematology and Oncology, Sofia
  - National Center of Haematology & Transfusiology, Sofia
  - Clinic of Haematology, Multiprofiled Hospital for Active Treatment "Sveta Marina", Varna
- Croatia (6):
  - Klinicki Bolnicki Centar Rijeka Interna Klinika, Rijeka
  - Klinika Bolnica SPLIT - Klinika za Unutarnje Bolesti, Split
  - KBC Zagreb - Klinika za Unutarnje Bolesti, Zagreb
  - Klinicka Bolnica "Dubrava" Klinika za Unutarnje Bolesti, Zagreb
  - Klinicka Bolnica "Sestre milosrdnice" Klinika za Unutarnje Bolesti, Zagreb
  - Klinicka Bolnica MERKUR - Klinika za Unutarnje Bolesti, Zagreb
- Czechia (6):
  - Interni Hemato-Onkologicka Klinika, Brno
  - Hematologicka Klinika, Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Onkologicke Centrum J.G. Mendela, Novi Jicin
  - Interni Klinika, Oddeleni Hematoonkologie, Olomouc
  - Interni Klinika, Oddeleni Hematoonkologie, Prague
  - Hematologicka Klinika, Fakultni Nemocnice Kralovske Vinohrady Srobarova, Prague
- France (3):
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - CHU de Nancy - Hopital Brabois, Nancy
  - Hematologie - CHU Purpan Place du Dr. Baylac, Toulouse
- Germany (15):
  - Charite, Universitatsmedizin Berlin, Campus Robert-Rossle Klinik, Berlin
  - Med. Klinik I/University Bonn, Bonn
  - Universitaetsklinik - Klinik fur innere Medizin, Cologne
  - Medizinische Klinik und Poliklinik I/Carl-Gustav-Carus University, Dresden
  - Hematology, Oncology & Clinical Immunology/Heinrich-Heine-University, Düsseldorf
  - Abt. Haematologie - Onkologie/ Allg. Krankenhaus, Hamburg
  - Allgemeinse Krankenhaus St. Georg Hamatologische Abteilung, Hamburg
  - Medizinische Klinik Abteilung Innere V/Universitatsklinikum, Heidelberg
  - Universitat Schleswig Holstein II Med. Klinik, Kiel
  - Medizinische Klinik und Poliklinik III/Klinikum der Universitaet Muenchen, München
  - Innere Medizin University Hospital, Münster
  - Abteilung Haematologie - Univeresitaetsklinikum, Saale
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart, Stuttgart
  - Universitaetsklinik - Abteilung Innere Medizin III, Ulm
  - Med. Klinik II/Klinikum of the Julius-Maximilians-University, Würzburg
- Hungary (4):
  - National Medical Centre Dpt Haematology, Budapest
  - Petz Aladar Megyei Oktato Korhaz, II. Belgyogyaszat, Győr
  - Pandy Kalman Megyei Korhaz, Megyei Onkologiai Centrum, Gyula
  - Szent-Gyorgyi Albert University II Clinic of Internal Medicine, Szeged
- India (9):
  - Nizam's Institute of Medical Sciences, Department of Medical Oncology, Hyderabaad
  - Department of Medical Oncology, Amrita Institute of Medical Sciences, Kerala
  - Orchid Nursing Home, Kolkata
  - Department of Medical Oncology, Dayanand Medical College DMCH, Ludhiana
  - Department of Medical Oncology/Tata Memorial Hospital, Mumbai
  - Department of Medical Oncology, S.L. Raheja Hospital, Mumbai
  - Department of Medical Oncology, Jaslok Hospital and Research Centre, Mumbai
  - Department of Medical Oncology, Deenanath Mangeshkar Hospital, Pune
  - Department of Medical Oncology/Regional Cancer Centre, Trivandrum
- Italy (2):
  - Instituto di Ematologia e Oncologia Medica, Bologna
  - Dipartimento Medicina ed Oncologia Sperimentale - Divisione Universitaria di Ematologia Azienda Ospedaliera S. Giovanni Battista, Torino
- Philippines (6):
  - Department of Internal Medicine - Baguio General Hospital & Medical Center, Baguio City
  - Chong Hua Hospital, Cebu City
  - Doctors Clinic Makati Medical Center, Makati City
  - University of Sto Tomas Hospital, Manila
  - Doctors Clinic - National Kidney & Transplant Institute, Quezon City
  - St. Luke's Medical Center, Quezon City
- Poland (10):
  - SPSK, Klinika Hematologii Akademii Medycznej, Bialystok
  - Klinika Hematologii Akademii Medycznej w Gdanskuul, Gdansk
  - Katedra i Klinika Hematologii i Transplantacji Szpiku - Slaska Akademia Medyczna, Katowice
  - Swietokrzyskie Centrum Onkologii SPZOZ Poradnia Hematologii, Kielce
  - Klinika Hematologii Uniwersytetu Medycznego, Lodz
  - Klinika Chorob Wewnetrznych i Hemagologii, Warsaw
  - Katedra i Klinika Hematologii, Onkologii I Chorob Wewnetrznych, Warsaw
  - Instytut Hematologii i Transfuzjologii - Klinika Hematologiczna, Warsaw
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Klinika Hematologii Nowotworow Krwi i Transplantacji - Szpiku Akademii Medycznej, Wroclaw
- Portugal (3):
  - Hospital da Universidade de Coimbra - Servico de Hematologia Clinica, Coimbra
  - Instituto Portugues de Oncologia, Lisbon
  - Hospital Geral de Santo Antonio - Servico de Hematologia Clinica, Porto
- Serbia (3):
  - Institute of Hematology, Clinical Centre of Serbia, Belgrade
  - Clinic for Hematology, Clinical Centre Nis, Niš
  - Clinic for Hematology, Clinical Centre Novi Sad, Novisad
- Slovakia (3):
  - Department of Internal Medicine, National Cancer Institute, Bratilslava
  - Hematology Department University Hospital, Bratilslava
  - Hematology Department, University Hospital PJS, Košice
- South Africa (6):
  - University of Free State, Faculty of Health Science, Dept of Hematology & Cell Biology, Bloemfontein
  - Tygerberg Hospital, University of Stellenbosch, Department of Haematology, Cape Town
  - Department of Haematology, UCT Medical School, Cape Town
  - Chris Hani Baragwanath Hospital, Clinical Haematology Unit, Johannesburg
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Johannesburg Hospital, Department of Medical Oncology, Parktown
- United Kingdom (4):
  - Oncology Research Unit Heartlands Hospital, Birmingham
  - Clinical Haematology, Guy's Hospital, London
  - Haematology Department - King's College Hospital, London
  - Department of Haematology-Oncology, The Royal Marsden NHS Foundation Trust, Surrey

REFERENCES:
- [Background] Kropff M, Baylon HG, Hillengass J, Robak T, Hajek R, Liebisch P, Goranov S, Hulin C, Blade J, Caravita T, Avet-Loiseau H, Moehler TM, Pattou C, Lucy L, Kueenburg E, Glasmacher A, Zerbib R, Facon T. Thalidomide versus dexamethasone for the treatment of relapsed and/or refractory multiple myeloma: results from OPTIMUM, a randomized trial. Haematologica. 2012 May;97(5):784-91. doi: 10.3324/haematol.2011.044271. Epub 2011 Dec 1. PMID 22133776
- [Background] Kropff M, et al. OPTIMUM Dose of Thalidomide for Relapsed Multiple Myeloma. Presented at American Society of Hematology 2009, New Orleans, LA. Abstract No. 959